CLINICAL TRIAL: NCT04745195
Title: Diagnostic and Risk Criteria for Complement Defects in Thrombotic Microangiopathy and Amplifying Conditions, Such as Severe Hypertension: The COMPETE Study.
Brief Title: Complement Prospective Evaluation of Thrombotic Microangiopathy on Endothelium
Acronym: COMPETE
Status: Recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Sjoerd Timmermans, Principal Investigator, Maastricht University Medical Center
Other Study IDs: NL74928.068.20; 23OK1056 (Other Grant/Funding Number: Dutch Kidney Foundation)
Record Dates: First submitted 2021-01-06; First posted 2021-02-09 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Thrombotic Microangiopathies; Hemolytic Uremic Syndrome, Atypical; Hemolytic-Uremic Syndrome
MeSH Terms: conditions — Thrombotic Microangiopathies; Atypical Hemolytic Uremic Syndrome; Hemolytic-Uremic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — The following samples will be obtained and stored at the time of presentation and during follow-up:
  * DNA
  * Kidney tissue sections (on indication)
  * Plasma
  * Serum
  * Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Complement-mediated thrombotic microangiopathy
- Thrombotic microangiopathty with normal complement regulation

SUMMARY:
Thrombotic microangiopathy (TMA) is a severe and life-threatening condition, often affecting the kidneys and brain. It can occur on the background of various clinical conditions. Dysregulation of the alternative pathway of complement may be the etiological factor and this type of TMA is classified, according to the current nomenclature, as primary atypical hemolytic uremic syndrome (HUS). Half the patients with primary atypical HUS present with rare variants in complement genes, although coexisting conditions are often needed for the TMA to become manifest. In patients with secondary atypical HUS, certain coexisting conditions appear to drive the disease and treatment should target the underlying condition to remit the TMA.

Recently, the investigators demonstrated, by using a novel in-house developed functional endothelial cell-based test, that complement dysregulation and overactivation is the dominant cause of disease and its sequelae in a subset of patients with secondary atypical HUS, having impact on treatment and prognosis. The investigators did first prove this concept in patients presenting with TMA and hypertensive emergency. A prospective study is needed to further corroborate these findings along the spectrum of TMA. The investigators hypothesize that their functional endothelial cell-based test, the so-called "HMEC" test, can better categorizes the TMA into different groups with potential therapeutic and prognostic implications. Thus, paving the road to the ultimate goal of precision medicine.

ELIGIBILITY:
Inclusion Criteria:

* Males or females at least 18 years of age;
* Have acute kidney injury, defined as estimated GFR <45 mL/min/1.73m2;
* Have documented TMA either on peripheral blood, defined as Coombs negative microangiopathic hemolytic anemia (hematocrit <30%, hemoglobin <6.5 mmol/L [<10 g/dL], lactate dehydrogenase >500 U/L, and either schistocytes on peripheral blood smear or undetectable haptoglobin), and platelets <150,000 per µL, or kidney biopsy;
* Have primary atypical HUS or a coexisting condition linked to complement dysregulation:

  * Hypertensive emergency, defined as SBP/DBP of >180/120 mmHg and impending organ damage secondary to hypertension (at least one of the following: neurologic disease, hypertensive retinopathy grade III and/or IV, left ventricular hypertrophy); OR
  * Pregnancy, including 12 weeks postpartum; OR
  * Kidney donor recipient; OR
  * Systemic auto-immune disease associated with TMA, including systemic sclerosis, systemic lupus erythematosus, anti-phospholipid syndrome;
* Have the ability to understand the requirements of the study, provide written informed consent, and comply with the study protocol procedures.

Exclusion Criteria:

* Have secondary causes of hypertensive emergency, including renovascular hypertension, Cushing syndrome, aldosteronism, pheochromocytoma, thyroid disease;
* Have a nephropathy not related to thrombosis on kidney biopsy;
* Have ADAMTS13 deficiency, defined as ADAMTS13 activity <10%;
* Have a positive stool culture for Shiga toxin producing bacteria;
* Have positive serologic test for viral infections, including HIV and CMV;
* Have a history of malignant disease, excluding non-melanoma skin cancer;
* Have a history of bone marrow or solid organ transplantation, excluding kidney transplantation;
* Received at least one of the following agents: chemotherapeutics, sirolimus, anti-VEGF agents;
* Have a history of recent past exposure to illicit drug(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of at least 18 years of age presenting with TMA, either on peripheral blood or kidney biopsy, will be recruited at the emergency departments of (regional) hospitals affiliated to the Limburg Renal Registry, Maastricht University Medical Center, Maastricht, NLD. Patients who meet the eligibility criteria will be included.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2021-08-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The prevalence of complement-mediated TMA along the spectrum of TMA | 1 year

SECONDARY OUTCOMES:
The diagnostic performance of the "HMEC" test for the diagnosis of complement-mediated TMA | 1 year
The dynamics of ex vivo C5b9 formation on the endothelium during the course of TMA | every month for up to 1 year
The dynamics of ex vivo C5b9 formation on the endothelium as compared to routine complement measures during the course of TMA | every month for up to 1 year
Composite kidney endpoint: 50% eGFR decline, chronic kidney disease stage G5, end-stage kidney disease | 1 year
  The diagnostic and prognostic value of pathologic features and chronicity indices on kidney biopsy at the time of presentation
composite TMA endopoint: TMA recurrence, end-stage kidney disease | 1 year
  The prognostic value of genetic variants in complement genes

CONTACTS AND LOCATIONS:
Overall Officials: Pieter van Paassen, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided